CLINICAL TRIAL: NCT00332631
Title: High-Dose N-Acetylcysteine in Cardiac Surgery Patients at High-Risk of Postoperative Renal Dysfunction.
Brief Title: High-Dose N-Acetylcysteine in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H2004/01899
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Cardiac Surgery and Cardiopulmonary Bypass
Keywords: Cardiac surgery,; Cardiopulmonary bypass,; Oxidative stress,; Acute renal dysfunction,; N-acetylcysteine
MeSH Terms: interventions — Acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine
Drug: Placebo

SUMMARY:
At least 14% of patients develop kidney failure after cardiac surgery. Although this kidney failure can usually be treated effectively, a longer stay in intensive care is often required. While many patients suffer no long term ill effects after developing post-operative kidney failure, some require long term kidney dialysis. The investigators also know that patients who develop post-operative kidney failure are much more likely to die before they leave hospital.

Why some people develop kidney failure after cardiac surgery is not known. However, doctors suspect that the process of cardiopulmonary bypass (where the functions of the heart and lungs are taken over by a machine during the operation, to allow the surgeon to operate) overactivates some of the same mechanisms the body uses to defend itself against severe infection. Many of the cell changes by which severe infection causes kidney failure also occur after cardiopulmonary bypass. One of the main overactive defence mechanisms is the release of highly toxic compounds derived from oxygen - a process called 'oxidative stress'.

Another well-known cause of oxidative stress is paracetamol (Panadol) overdose. In large doses the oxidative stress caused by paracetamol damages cells in the liver, where it is digested, and the kidney. N-acetylcysteine is a drug in common use for the treatment of paracetamol overdose. Patients who would otherwise die of liver failure are routinely saved by N-acetylcysteine, which acts as a strong anti-oxidant.

The investigators believe that N-acetylcysteine might similarly reduce the oxidative stress which occurs during cardiac surgery, and so prevent or decrease the kidney failure which occurs in many patients. The investigators hope to give N-acetylcysteine (in similar doses to those used safely for paracetamol poisoning) to patients during, and for a day after cardiac surgery, and compare the effects with patients who have not had N-acetylcysteine. The drug, or a 5% glucose placebo, will be given through the drip which is present in all cardiac surgery patients. Whether a particular patient receives the drug or placebo will be decided at random, and neither the patient nor the investigators will know which has been given. The investigators will measure kidney function before and after the operation using the standard tests which are performed for the purposes of clinical care of every patient. Also, the investigators will do an extra test involving the collection of urine (from the urinary catheter every patient has after cardiac surgery), which provides an even better measure of kidney function. This is a potential benefit to the patient, as while this test is not routinely performed, the results will be available to the doctors in the intensive care unit. The investigators will also take four 20ml samples of blood, spaced before, during, and after the operation, from the arterial catheter routinely inserted in every patient. This is an insignificant amount of blood compared to that taken for other tests, and would have no adverse effects. This blood would be used to measure oxidative stress, and also some of the proteins inside the blood cells which are responsible for creating the toxic oxygen compounds. In this way the investigators will discover not only the effect of N-acetylcysteine, but the mechanism of that effect.

N-acetylcysteine is routinely used to treat paracetamol overdose with few side effects. An itchy skin rash is the only common side effect. Sometimes patients develop nausea and vomiting, but the treatment for this is usually very effective, and the drug will be stopped if it occurs. Rarely, as with all drugs, allergic reactions have been reported, but there are no other reported adverse effects.

There will be no extra risk to a patient who participates in the study, and no discomfort other than that normally associated with cardiac surgery. The itchy rash which occasionally develops with N-acetylcysteine would occur under anaesthetic, and would almost certainly be gone by the time the patient wakes up.

Informed consent will be obtained from the patient prior to the operation by one of the investigators or the ICU research nurse.

DETAILED DESCRIPTION:
Background

Renal impairment following cardiopulmonary bypass is common. 11.4% (1) to 42% (2) of patients with previously normal renal function show a postoperative rise in serum creatinine. While most of these patients do not require either short or long term renal replacement, the mortality of patients with acute renal failure is substantially greater than those who do not develop renal dysfunction1.

Cardiopulmonary bypass activates components of the non-specific immune system, which leads to the generation of compounds containing oxygen free radicals. A study of 14 patients undergoing cardiac surgery found increased levels of serum lipid peroxidation products (thiobarbituric acid reactive substances) within 15 minutes of the commencement of cardiopulmonary bypass, which returned to preoperative levels by the following morning. The total serum antioxidative capacity was correspondingly decreased intraoperatively, and remained decreased at 24 hours postoperatively (3). A similar study of total plasma antioxidant status showed decreased levels up to 72 hours postoperatively(4). It is clear that cardiopulmonary bypass causes oxidative stress and depletion of antioxidant capacity.

N-acetylcysteine is routinely used in the treatment of paracetamol overdose. Paracetamol is metabolised by the liver by cytochrome p450 to form a toxic reactive oxygen compound. This metabolite is normally detoxified by conjugation with hepatic reduced glutathione (GSH). In overdose, the GSH stores are depleted, leading to liver cell necrosis through oxidative damage. N-acetylcysteine is a sulfydryl group donor, which allows regeneration of GSH, thus augmenting the antioxidant defence of the liver. Treatment of paracetamol overdose is currently the only approved indication for N-acetylcysteine. Possible adverse reactions include an urticarial rash, nausea and vomiting, and an anaphylactoid reaction (involving hypotension, tachycardia, bronchospasm, and facial oedema). These reactions occur most commonly either during, or at the end of, the period of the loading dose infusion, and may be concentration related (5).

Oxidative stress can be produced experimentally using hypertonic glycerol. Intramuscular injection of hypertonic glycerol in rats precipitated acute renal failure associated with a marked decrease in renal reduced glutathione (GSH) levels. Pretreatment with N-acetylcysteine largely prevented these changes (6). During reperfusion after renal ischaemia in rats, renal blood flow was reduced compared to pre-ischaemic values. GFR was also reduced, and plasma peroxynitrite (a marker of nitric oxide synthesis, a component of oxidative stress) was increased. Pretreatment with N-acetylcysteine partially prevented these changes (7). N-acetylcysteine (combined with a nitric oxide donor and an endothelin converting enzyme inhibitor) also decreased the effect of renal ischaemia/reperfusion injury in dogs, in terms of improved renal function as well as reduced interstitial pro-inflammatory cytokines and inducible nitric oxide synthase (8).

Radiocontrast commonly causes renal dysfunction, in part through oxidative stress in the kidney. While not an approved indication, intravenous N-acetylcysteine has been used successfully to attenuate radiocontrast induced nephropathy, and was more effective than standard intravenous fluid prophylaxis (relative risk 0.28) (9). While not an approved product indication, N-acetylcysteine is currently used in our hospital for this purpose.

Infrarenal abdominal aortic aneurysm repair commonly causes ischaemia/reperfusion injury to the kidney, producing a similar oxidative stress to that of radiocontrast. A mixture of antioxidants including N-acetylcysteine given to patients undergoing infrarenal abdominal aortic aneurysm repair produced a significantly better creatinine clearance (compared to placebo controls) 48 hours postoperatively (10).

While never investigated for its effects on renal function after cardiac surgery, the effect of perioperative N-acetylcysteine on other systems has been studied. The oxidative burst response of neutrophils from patients undergoing cardiopulmonary bypass was significantly attenuated by infusion of N-acetylcysteine into the bypass circuit (11).

A study of dogs undergoing cardiopulmonary bypass found preload-recruitable stroke work was maintained at pre-bypass levels in those animals given N-acetylcysteine, whereas it fell in control animals. N-acetylcysteine significantly enhanced myocardial oedema resolution, and prevented the rise in plasma 8-isoprostane (a marker of oxidative stress) seen in control animals (12). Similar results were found in a study of 40 patients undergoing cardiac surgery: left ventricular biopsy specimens showed less 8-isoprostane content and less nitrotyrosine (a marker of nitric oxide production; nitric oxide can act as an oxygen free radical). There were no differences in haemodynamics or clinical outcomes noted, but unfortunately indices of renal function were not examined in this study (13).

Ascorbate is an antioxidant which might be expected to have a similar action to N-acetylcysteine. Supplemental ascorbate was given to 43 patients before, and for 5 days after, coronary artery bypass surgery. Patients receiving ascorbate had a 16.3% incidence of postoperative AF, compared to 34.9% in control subjects, perhaps by reducing oxidative damage to the myocardium (14).

Pulmonary endothelium-dependent vasodilation is usually impaired after cardiopulmonary bypass, a process thought to be related to reactive oxygen species. Pulmonary vasodilation induced by acetylcholine following cardiopulmonary bypass was better maintained in 12 patients given a cocktail of antioxidants (including N-acetylcysteine) compared to that in 10 control patients (15).

There is thus evidence that in the immune, cardiovascular and respiratory systems, N-acetylcysteine may be of benefit to patients undergoing cardiac surgery.

Clinical sepsis or experimental exposure to lipopolysaccharide stimulate cells of the inflammatory system to form oxygen free radicals. N-acetylcysteine decreases cytokine and adhesion molecule gene expression and NF-kB activation in vitro. In animal models of sepsis N-acetylcysteine reduces inflammatory cell chemotaxis and improves survival (as reviewed by ref. 16). In patients suffering oxidative stress due to sepsis, N-acetylcysteine results in decreased NF-kB activation and decreased IL-8 production (16).

Hypotheses N-acetylcysteine administered from the time of induction of anaesthesia prior to cardiac surgery and for 24 hours postoperatively results in decreased change in serum creatinine from baseline to peak level within first 5 postoperative days.

Other secondary outcomes which will be measured include:

* better creatinine clearance over the first postoperative day;
* shorter ICU stay;
* shorter hospital stay;
* lower serum creatinine levels on day 2 post-op;
* greater plasma antioxidant activity;
* less oxidative stress;
* less NF-kB activation in the cellular components of blood;
* less pro-inflammatory cytokine response; and
* less activation of the nitric oxide synthase pathway.

Study Design - overview and rationale

Patients will be randomised to receive N-acetylcysteine from the induction of anaesthesia until 24 hours postoperatively, or a placebo (5% glucose).

Serum creatinine is the most commonly used clinical indicator of renal function along with urine output. Both will be measured for 48 hours postoperatively - the time period during which renal impairment is most likely to develop. A more sensitive indicator of renal dysfunction is creatinine clearance. This will be measured over the first 24 hours postoperatively, and will form the primary end point of the study. As patients in our intensive care unit are routinely given frusemide to maintain a postoperative urine output of >0.5ml/kg/hr (once fluid volume, inotropy and vascular tone have been manipulated into what is judged to be acceptable ranges), the dose of frusemide required is also an indicator of renal function. Rarely are other diuretics given, though where this is the case it will also be noted.

The efficacy of N-acetylcysteine in preventing oxidative stress will be assessed using a measure of total plasma antioxidant activity (the bathocuproine assay) (17) and by quantification of the 8-isoprostane levels (18). Total antioxidant activity and 8-isoprostane have previously been shown to be affected by cardiac surgery and N-acetylcysteine.

Any renal effect of N-acetylcysteine will be correlated with levels of plasma pro-inflammatory cytokines (IL-1, IL-6 and TNF-alpha), which are known to be associated with oxidative-stress induced renal failure (19, 20). Activation of inducible nitric oxide production is also associated with renal failure (21), and the effect of N-acetylcysteine on nitric oxide synthase mRNA expression in the cellular components of blood will be assayed by real-time PCR. Nitric oxide production will be assessed by measurement of by plasma nitrotyrosine concentration. Assay of nitrotyrosine is superior to the traditional Greiss reaction (which measures nitrate and nitrite derivatives of nitric oxide), as nitrate and nitrite undergo renal excretion, and many of these patients will have altered renal function.

At a molecular level, many of the genes responsible for stimulating oxidative stress are regulated by the promoter NF-kB. The cellular components of blood will be assayed for NF-kB using an established ELISA technique (22) thought to be more sensitive than the electrophoretic mobility shift assay used to demonstrate an effect of N-acetylcysteine in human sepsis (16). NF-kB in the cellular components of blood will also be assayed using real-time PCR.

Randomisation The randomisation will be based on random numbers generated by computer. Once consent is obtained, the allocation of either treatment with N-acetylcysteine or placebo will be organised by an independent person (clinical trials pharmacist) who will dispense the coded infusion bags. This will be delivered to the anaesthetic staff looking after the patient in theatre, and the ICU nurse caring for the patient postoperatively.

Detailed protocol Immediately following the induction of anaesthesia, prior to the first surgical incision, N-acetylcysteine will be administered in a dose of 150 mg/kg IV in 200 mL 5% glucose over 15 minutes followed by continuous IV infusion of 50 mg/kg in 500 mL 5% glucose over 4 hours, then 100 mg/kg in 1 L 5% glucose over 20 hours (total dose 300 mg/kg in 24 hours). This is the standard dose of N-acetylcysteine used clinically in paracetamol overdose (5.) Patients randomised to receive placebo will receive an equivalent volume of 5% glucose. The appearance of the 5% glucose and N-acetylcysteine solutions is similar, and there will be no marking on the infusion bag other than an identifying study number.

A 24 hour urine collection will begin immediately on arrival in ICU, to allow determination of creatinine clearance. This will be measured in the hospital clinical pathology laboratory. Creatinine clearance will be the primary endpoint of the study.

Clinical data will be recorded as detailed below by the investigators or the ICU research nurse.

Four 20 ml samples of heparinised blood will be taken from the arterial line for cytokine and molecular analysis. Samples will be taken immediately after the induction of anaesthesia, on arrival in the intensive care unit, and 6 and 24 hours postoperatively. Immediately following collection, the blood will be centrifuged at low speed to separate the plasma from the cellular components, both of which will be stored in aliquots at -70 degrees prior to batch analysis.

Analysis of plasma total antioxidant activity and 8-isoprostane, IL-1, IL-6, TNF-alpha and nitrotyrosine concentrations will be performed using commercially available ELISA reagent kits (Oxford Biomedical Research, Oxis Research, BioCore). The cellular components of blood will be assayed for NF-kB concentration using a commercially available ELISA kit (Oxford Biomedical Research), and for iNOS and NF-kB mRNAs using a real-time PCR machine and Applied Biosystems pre-developed assay reagents with 18S as the endogenous control. The principal investigator has experience of these or similar techniques.

Statistics and power calculation Using data available from our cardiac surgery database of over 2500 patients in the last 5 years, we expect a mean increase in serum creatinine from baseline to a peak value of 50 micromol/L in the control group, with a standard deviation of 30 micromol/L. Given these changes, 60 patients are needed to have a 90% power of detecting a 30 micromol/L difference between the control and the intervention group at an alpha of 0.05.

Data collection Data collection will be performed by the principal investigator, ICU research nurse and ICU nursing staff.

The following variables will be obtained:

Name gender, age, and medical record number Date of admission to ICU Operative procedure and time on cardiopulmonary bypass Preoperative assessment of left ventricular function Serum creatinine and urea preoperatively, immediately postoperatively, and every 24 hours thereafter (as measured for clinical purposes) Doses of frusemide administered (or rate of frusemide infusion) Use of inotropes Cardiac output whenever measured for clinical purposes in the first 24 hours postoperatively Urine output in each 6 hour period for the 24 hours postoperatively Date of discharge from ICU and hospital or death

Protocol violations All protocol violations will be recorded. It will then be decided whether the nature of such violation had been such that the patient should be excluded from primary data analysis. Such evaluation will be blinded to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age above 70 years
* Preexisting renal impairment (preoperative serum creatinine level >120µmol/L
* New York Heart Association class III/IV or Moderate to poor left ventricular dysfunction
* Valve surgery or complex cardiac surgery
* Redo cardiac surgery
* Insulin-dependent diabetes mellitus

Exclusion Criteria:

* Age <18 years
* Known allergy or hypersensitivity to N-acetylcysteine
* Emergency cardiac surgery
* Planned off-pump cardiac surgery
* Enrolled in conflicting research study
* Known blood-borne infectious disease
* Chronic inflammatory disease on immunosuppression
* Chronic moderate to high dose corticosteroid therapy (>10mg/d prednisone or equivalent)
* End stage renal disease (serum creatinine >300µmol/L)
* Patients receiving pre-op IV nitrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2006-03

PRIMARY OUTCOMES:
Absolute change in serum creatinine from baseline to peak level within the first five postoperative days.

SECONDARY OUTCOMES:
Relative change in serum creatinine,
Highest serum creatinine,
Change in estimated glomerular filtration rate (eGFR),
Change in serum cystatin C (as a serum creatinine-independent marker of renal function during and after NAC administration (Hoffmann et al. JASN 2004),
Urinary output
Use of renal replacement therapy (RRT)
Acute renal dysfunction
Duration of ventilation,
Chest tube drainage,
Need for return to operating room,
Incidence of post-operative atrial fibrillation (AF),
Duration of stay in the intensive care unit (ICU)
Duration of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD, FRACP, Principal Investigator — Austin Health
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Haase M, Haase-Fielitz A, Ratnaike S, Reade MC, Bagshaw SM, Morgera S, Dragun D, Bellomo R. N-Acetylcysteine does not artifactually lower plasma creatinine concentration. Nephrol Dial Transplant. 2008 May;23(5):1581-7. doi: 10.1093/ndt/gfm818. Epub 2008 Jan 17. PMID 18202091